CLINICAL TRIAL: NCT04591171
Title: Assessing the Feasibility of N-of-1 Trials in Children With Hypertension and Chronic Kidney Disease: a Pilot Study
Brief Title: Assessing the Feasibility of N-of-1 Trials in Children With Hypertension and Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Children's Hospital of Philadelphia (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joyce Philip Samuel, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-20-1005
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Hypertension; Chronic Kidney Diseases
Keywords: n-of-1 trial
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- n-of-1 trial guided clinical decision making (Experimental)
  Interventions: Procedure: n-of-1 trial guided clinical decision making

INTERVENTIONS:
Procedure: n-of-1 trial guided clinical decision making — The n-of-1 trial will, on the level of the individual patient, test which treatment strategy produces superior blood pressure reduction without unacceptable side effects. After discussion with the patient/caregiver dyad to identify whether they have specific concerns about particular medications, the nephrologist (clinician) will decide which two drugs and dosages will be tested in the n-of-1 trial (the protocol does not determine drug or dose). The two drugs chosen by the clinician will be assessed at clinician-selected dosing in a randomized treatment order (e.g., ABAB) for two weeks per treatment period and two treatment periods per drug.

SUMMARY:
The purpose of this study to test whether n-of-1 trial-guided clinical decision-making improves blood pressure control in hypertensive children with chronic kidney disease (CKD) and end-stage renal disease (ESRD).

ELIGIBILITY:
Inclusion Criteria:

* hypertension
* CKD stage 2-5
* requiring antihypertensive medication per clinician judgement.

Exclusion Criteria:

* renal transplant anticipated or occurred within 6 months of screening
* transfer out of our practice setting anticipated within 6 months
* unable to complete 24 hour arterial blood pressure monitoring (ABPM) due to developmental or behavioral limitations

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce P Samuel, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas at Houston Medical School; Pediatric Nephrology and Hypertension Clinics, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-of-1 Trial Guided Clinical Decision Making
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | N-of-1 Trial Guided Clinical Decision Making
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 11 [6 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Transplant or Dialysis Status [Count of Participants; unit: Participants]
  Transplant | 4
  Dialysis | 0
  non-dialysis CKD | 5
distance from home to clinic [Median (Full Range); unit: miles] | 30 [15 to 99]
glomerular filtration rate (GFR) [Mean (Full Range); unit: mL/min/1.73m^2] | 65 [19 to 105]

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hour Mean Arterial Pressure (MAP)
Description: 24-hour mean arterial pressure (MAP) is the mean arterial pressure over 24 hours [ambulatory blood pressure monitoring (ABPM) will be used to record blood pressure every 20 min for 24 hours, and all recordings will be averaged to obtain 24-hour MAP]. 24-hour MAP will be assessed at baseline and at 6 months, and the change between baseline and 6-months will be reported.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | N-of-1 Trial Guided Clinical Decision Making
Number analyzed (Participants) | 9
mmHg | 1.4 (5.9)

2. Secondary Outcome: Number of Participants With Target Blood Pressure
Description: Target blood pressure is 24-hour mean arterial pressure (MAP) at less than the 50th percentile.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-of-1 Trial Guided Clinical Decision Making
Number analyzed (Participants) | 9
Participants | 4

3. Secondary Outcome: Number of Participants With Target Blood Pressure
Description: Target blood pressure is 24-hour mean arterial pressure (MAP) at less than the 50th percentile.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | N-of-1 Trial Guided Clinical Decision Making
Number analyzed (Participants) | 9
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | N-of-1 Trial Guided Clinical Decision Making
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04591171/Prot_SAP_000.pdf